CLINICAL TRIAL: NCT05891808
Title: Expression of miR-155 in Migraine: Association With Different Phenotypes and Disease Severity
Brief Title: miR-155 Expression in Episodic and Chronic Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: miRNA-155 - MiG
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Migraine; Headache; Pain; Chronic Migraine
Keywords: MicroRNA; miR-155; Peripheral blood mononuclear cells; Monocytes
MeSH Terms: conditions — Migraine Disorders; Headache; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Healthy subjects without present or past history of headache according to ICHD-III criteria.
- Episodic Migraine: Patients with a diagnosis of migraine without or with aura, with episodic pattern, according to ICHD-III criteria.
- Chronic Migraine: Patients with a diagnosis of chronic migraine with or without medication overuse headache according to ICHD-III criteria.

SUMMARY:
Migraine is a common, yet often disabling, neurological disease that affects over 1 billion people around the world. It's the second most disabling disease globally and the leading cause of disability for people under the age of 50, especially women. The effects of migraine aren't limited to the individual, with a tremendous economic impact on families, friends, and employers. To help reduce this burden, research is now focusing on developing biomarkers that can help with diagnosis, predicting response to treatments, and identifying those at risk of developing chronic migraine.

MicroRNAs (miRNAs) are one of the most promising classes, as they can modulate gene expression and affect a wide range of cellular processes. Other studies have already observed different miRNA expression in those with episodic migraine or chronic migraine, but no specific miRNAs have been identified as a strong and specific migraine signature. miRNA-155 is of particular interest, as it has been linked to inflammation and pain, and may be a potential target for migraine treatments.

It is known that the immune system plays a role in migraine headaches. Monocytes, a type of immune cell, may be involved in the development of migraines. Certain medicines, such as aspirin, can affect monocyte function and have been used to treat migraines. Recent research has also shown that microRNAs can regulate the activity of these cells and influence inflammation, which may be linked to migraine attacks.

This study aims to investigate the role of miRNA-155 and monocyte differentiation in migraine patients, and in particular its association with migraine phenotype and severity. We aim to study three groups of subjects: Episodic migraine (EM), Chronic migraine with or without Medication Overuse Headache (CM-MOH) and Healthy Controls (HCs).

DETAILED DESCRIPTION:
Background:

Depending on the median frequency of headache, migraine is defined as episodic migraine (EM) (for those who have less than 15 migraine days per month), or chronic migraine (for those who have at least 15 headache days per month, 8 of which with migraine features, for at least three months). The chronification of migraine is often associated with a progressive increase of acute medications intake, leading to a condition known as Medication Overuse Headache (CM-MOH).

So far, there are no validated and reliable biomarkers of migraine, but the headache scientific community is intensely investigating the neurobiological signatures of migraine. Validated biological biomarkers may allow several steps forward in the management of migraine by: (I) refining the diagnosis according to biological features; (II) predicting the response to advanced therapies; (III) predicting which patients are at the greatest risk of migraine chronification and mark different phases of the migraine cycle; (IV) the identification of novel molecular targets for drugs development. Fulfilling these purposes, a class of molecules that has recently gained enormous interest are microRNAs (miRNAs). miRNAs are small endogenous noncoding RNAs that are around 22 nucleotides in length. miRNAs operate as post-transcriptional regulator of gene expression by promoting messenger RNA (mRNA) degradation or repressing mRNA translation. The regulation process performed by miRNAs is complex and articulated since an individual miRNA might target hundreds of different mRNAs, and conversely, each mRNA may be regulated by multiple miRNAs. It has been estimated that more than 60% of all protein-coding genes are regulated by miRNAs which consequentially determine the pleiotropic modulation of a wide variety of cellular processes involving differentiation, development and signaling. miRNAs are involved in the generation and maintenance of pain and several evidence suggest that specific miRNAs could play a role in migraine.

The micro-MIG study corroborated the hypothesis that different miRNAs expression is altered in EM and CM when compared to a control group, although no specific miRNAs were identified as a strong and specific migraine molecular signature.

miRNA-155 can be considered as a master regulator of inflammation since its expression can modulate many inflammatory stimuli such as: interleukin 1β (IL-1β), tumor necrosis factor alpha (TNF-α), alarmins (eg, IL-1α), hypoxia, nuclear factor erythroid 2-related factor 2 (NRF2), pathogen-associated and damage-associated molecular patterns as well as to toll-like receptor ligand (TLR) in various cell types. Recently, several lines of preclinical evidence further highlighted the role of miRNA-155 in inflammation and pain generation and maintenance also as a feasible therapeutic target. The inhibition of miRNA-155 can alleviate hyperalgesia and bone cancer pain as well as neuropathic pain in in-vivo rodent models. Therefore, it can be inferred that miRNA-155 might also play an important role in neurogenic inflammation, a process supposed to take place in the trigeminovascular system, and related to the pathogenic mechanisms underlying migraine pain.

Monocytes are immune system components which may play a role in migraine. For example, abortive migraine treatment may influence monocyte function. Acetylsalicylic acid inhibits monocyte chemotaxis, whereas metoprolol, metoclopramide, dihydroergotamine, and sumatriptan have no impact. microRNAs have been shown to regulate macrophage polarization and subsequent effects on inflammation.

Aims:

In order to shed light upon the mediators involved in migraine pathophysiology and its chronification, we aim to asses the different expression of miRNA-155 (in monocytes) in patients with EM, CM-MOH and healthy controls (HCs). Secondly, we aim to provide information about distribution of monocyte phenotype in the three groups.

Expected evaluations:

For all patients is scheduled a single evaluation over time - baseline (T0) - in the interictal migraine phase, during which they will undergo:

* informed consent signing
* screening visit
* clinical and demographic data collection (based on revision of a headache diary)
* venous blood sampling All patients will be evaluated in the morning, after night fasting, and in the inter-ictal migraine phase.

Detailed description of the methods planned for the biochemical analyses could be found here:

* 10.1186/s10194-020-01189-0;
* 10.1177/0333102420949201.

Sample size calculation:

Sample size was calculated from preliminary data available, which showed a difference in miR-155 levels in peripheral mononuclear cells of 1.69 RQ (relative quantification), with standard deviations of 1.15, and 2.69 RQ in healthy control and episodic migraine subjects, respectively. This difference has been assumed the same between episodic and chronic subjects.

Therefore, assuming a statistical power of 80 percent, a significance level of 95 percent and performing Bonferroni correction, we need a sample size of 24 subjects for the three experimental groups (HCs, CM-MOH and EM). Considering possible variability in dosing, we will enroll at least 30 subjects per group.

Pre-planned statistical analysis:

The difference between of miR155 expression among CM-MOH, EM and HCs will be determined by parametric (ANOVA) or non-parametric (Kruskal-Wallis) tests depending on the distribution of data. Parametric or non-parametric correlations will be used to measure the relationship between biochemical variables and clinical variables in CM-MOH and EM patients. Multivariate analyses will be performed according to the results of the univariate analysis. Statistical significance will be set at the 5% level (p<0.05).

ELIGIBILITY:
Healthy Controls:

Inclusion Criteria:

1. age between >18 and <65 years, of both genders

Exclusion criteria:

1. diagnosis of primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension type headache is allowed)
2. diagnosis of neurological disorders
3. diagnosis of medical conditions considered clinically relevant by the researcher
4. pregnant and lactating women
5. taking NSAIDs, triptans or opiates in the previous 24 hours

Episodic Migraine

Inclusion Criteria:

1. diagnosis of migraine without or with aura according to ICHD-III criteria
2. age between >18 and <65 years of both genders
3. have completed a headache diary for at least 3 months at the time of enrollment

Exclusion criteria:

1. history of chronic migraine or other chronic headache subtypes according to ICHD-III criteria
2. concomitant diagnosis of other primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension headache is allowed)
3. diagnosis of other neurological disorders
4. diagnosis of medical conditions considered clinically relevant by the researcher
5. diagnosis of chronic pain syndrome of any nature
6. pregnant and lactating women
7. use of substances of abuse
8. taking NSAIDs, triptans or opiates in the previous 24 hours

Chronic Migraine

Inclusion Criteria:

1. diagnosis of chronic migraine with or without concomitant diagnosis of medication overuse headache according to ICHD-III criteria
2. history of chronic migraine for at least 1 year
3. age between >18 and <65 years, of both sexes
4. have completed a headache diary for at least 3 months at the time of enrollment

Exclusion criteria:

1. concomitant diagnosis of other primary and/or secondary headache according to ICHD-III criteria (only diagnosis of sporadic tension headache is allowed)
2. concomitant diagnosis of other neurological disorders
3. diagnosis of medical conditions considered clinically relevant by the researcher
4. diagnosis of chronic pain syndrome of any nature
5. pregnant and lactating women
6. use of substances of abuse
7. taking NSAIDs, triptans or opiates within the previous 24 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to enroll a representative population of patients affected by EM and CM-MOH. All patients will be consecutively enrolled among those attending the clinics of the Headache Science Center of the IRCCS Mondino Foundation of Pavia (Italy).
  A set of healthy controls, without a diagnosis of present or past headache, will be enrolled as control group.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of miR-155 expression in peripheral monocytes between the three study groups: chronic migraine, episodic migraine and healthy control. | Baseline (T0).
  miRNA-155 gene expression will be evaluated by real-time reverse transcription (RT-PCR). This assessment will be then normalized with U6 (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ).

SECONDARY OUTCOMES:
Cytofluorimetric evaluation of monocytes to determine their phenotype and subtype and the different colocalization of these between the three study groups: chronic migraine, episodic migraine and healthy control. | Baseline (T0).
  Phenotype evaluation: Cytofluorimetric assessment of the percentage of classical and non-classical M1 inflammatory (CD80+), and classical and non-classical M2 anti-inflammatory (CD163+) monocytes.
  Classical monocytes are characterized by high level expression of the CD14 cell surface receptor (CD14++ CD16- monocyte). Non-classical monocyte show low level expression of CD14 and additional co-expression of the CD16 receptor (CD14+CD16++ monocyte).
Comparison of gene expression in peripheral monocytes of pro-inflammatory (IL-1B, TNF-alpha) and anti-inflammatory (IL-10) cytokines between the three study groups: chronic migraine, episodic migraine and healthy control. | Baseline (T0).
  Cytokines genes expression will be evaluated by real-time reverse transcription (RT-PCR). This assessment will be then normalized with UBC (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ).
Comparison of miR-382-5p and miR-34a-5p expressions in peripheral monocytes between the three study groups: chronic migraine, episodic migraine and healthy control. | Baseline (T0).
  miR-382-5p and miR-34a-5p expressions will be evaluated by real-time reverse transcription (RT-PCR). This assessment will be then normalized with U6 (a type of small nuclear RNA used as housekeeping gene) and expressed as Relative Quantification (RQ).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

REFERENCES:
- [Background] Essandoh K, Li Y, Huo J, Fan GC. MiRNA-Mediated Macrophage Polarization and its Potential Role in the Regulation of Inflammatory Response. Shock. 2016 Aug;46(2):122-31. doi: 10.1097/SHK.0000000000000604. PMID 26954942
- [Background] Yamanaka G, Suzuki S, Morishita N, Takeshita M, Kanou K, Takamatsu T, Suzuki S, Morichi S, Watanabe Y, Ishida Y, Go S, Oana S, Kashiwagi Y, Kawashima H. Role of Neuroinflammation and Blood-Brain Barrier Permutability on Migraine. Int J Mol Sci. 2021 Aug 19;22(16):8929. doi: 10.3390/ijms22168929. PMID 34445635
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Ashina M, Terwindt GM, Al-Karagholi MA, de Boer I, Lee MJ, Hay DL, Schulte LH, Hadjikhani N, Sinclair AJ, Ashina H, Schwedt TJ, Goadsby PJ. Migraine: disease characterisation, biomarkers, and precision medicine. Lancet. 2021 Apr 17;397(10283):1496-1504. doi: 10.1016/S0140-6736(20)32162-0. Epub 2021 Mar 25. PMID 33773610
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Gazerani P. Current Evidence on Potential Uses of MicroRNA Biomarkers for Migraine: From Diagnosis to Treatment. Mol Diagn Ther. 2019 Dec;23(6):681-694. doi: 10.1007/s40291-019-00428-8. PMID 31612314
- [Background] Gallardo VJ, Gomez-Galvan JB, Asskour L, Torres-Ferrus M, Alpuente A, Caronna E, Pozo-Rosich P. A study of differential microRNA expression profile in migraine: the microMIG exploratory study. J Headache Pain. 2023 Feb 17;24(1):11. doi: 10.1186/s10194-023-01542-z. PMID 36797674
- [Derived] Greco R, Bighiani F, Demartini C, Zanaboni A, Francavilla M, Facchetti S, Sproviero D, Vaghi G, Allena M, Martinelli D, Corrado M, Guaschino E, Ghiotto N, Bottiroli S, Cammarota F, Antoniazzi A, Grillo V, Sances G, Tassorelli C, De Icco R. miR-382-5p and miR-34a in migraine: Expression in monocytes and a post-hoc exploratory comparison with expression in peripheral blood mononuclear cells. Cephalalgia. 2025 Dec;45(12):3331024251386769. doi: 10.1177/03331024251386769. Epub 2025 Dec 4. PMID 41342643
- [Derived] Greco R, Bighiani F, Demartini C, Zanaboni A, Francavilla M, Facchetti S, Vaghi G, Allena M, Martinelli D, Guaschino E, Ghiotto N, Bottiroli S, Corrado M, Cammarota F, Antoniazzi A, Mazzotta E, Pocora MM, Grillo V, Sances G, Tassorelli C, De Icco R. Expression of miR-155 in monocytes of people with migraine: association with phenotype, disease severity and inflammatory profile. J Headache Pain. 2024 Aug 27;25(1):138. doi: 10.1186/s10194-024-01842-y. PMID 39187749